CLINICAL TRIAL: NCT06038942
Title: The Acceptability and Effectiveness of Formal Versus Informal Mindfulness Instruction Among University Students With Self-reported ADHD, Lived Experience of Nonsuicidal Self-injury, or Stress: An Online Randomized Controlled Trial
Brief Title: Formal Versus Informal Mindfulness Among University Students With Self-reported ADHD, Nonsuicidal Self-injury, or Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Concordia University, Montreal (Other); University of Ottawa (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-06-016
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Nonsuicidal Self-injury; ADHD; Mindfulness
Keywords: nonsuicidal self-injury; ADHD; formal mindfulness; informal mindfulness; university students
MeSH Terms: conditions — Self-Injurious Behavior; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formal mindfulness instruction (Experimental)
  Interventions: Behavioral: Formal mindfulness instruction
- Informal mindfulness instruction (Experimental)
  Interventions: Behavioral: Informal mindfulness instruction
- Inactive control (No Intervention): An equal number of university students from all groups will participate in this arm (i.e., those with ADHD, those with a history of nonsuicidal self-injury, and those with self-reported stress). Participants assigned to the inactive control condition will not complete any tasks during the four-week intervention period.

INTERVENTIONS:
Behavioral: Formal mindfulness instruction — An equal number of university students from all groups will participate in this arm (i.e., those with ADHD, those with a history of nonsuicidal self-injury, and those with self-reported stress). The formal mindfulness instruction will consist of four weekly 1 hour-long group sessions, held on Webex (i.e., online) over four consecutive weeks. Participants will learn foundational principles around the role of mindfulness in relation to emotion regulation, stress, and self-compassion.
  They will also be taught formal mindfulness practices (e.g., sitting meditation, body scan, thought meditation, loving-kindness meditation) during the group sessions and will be asked to commit to practicing the strategies independently throughout the project period.
  Arms: Formal mindfulness instruction
Behavioral: Informal mindfulness instruction — An equal number of university students from all groups will participate in this arm (i.e., those with ADHD, those with a history of nonsuicidal self-injury, and those with self-reported stress). The informal mindfulness instruction will consist of four weekly 1 hour-long group sessions, held on Webex (i.e., online) over four consecutive weeks. Participants will learn foundational principles around the role of mindfulness in relation to emotion regulation, stress, and self-compassion.
  They will also be taught how to integrate informal mindfulness into their daily routine and will be guided through a series of demonstrations within the group sessions. Participants will be asked to commit to practicing informal mindfulness independently throughout the project period.
  Arms: Informal mindfulness instruction

SUMMARY:
The present study will use a randomized controlled design to investigate group differences between university students with self-reported stress (comparison group), ADHD, or a history of nonsuicidal self-injury (NSSI) in response to a four-week mindfulness instruction program across conditions (formal mindfulness program, informal mindfulness program, inactive control) in terms of the intervention's acceptability and effectiveness.

DETAILED DESCRIPTION:
As post-secondary students report increasing levels of stress and difficulty coping with the challenges of university, student services have had to consider alternative approaches to meet the demand for student support. Thus, there has been a move towards extending support beyond traditional mental health services to include the teaching of resilience-building strategies. These resilience-building activities use pedagogical principles and are commonly instructional programs offered to groups of students. These programs often use mindfulness (i.e., purposeful attention to the present moment with nonjudgmental acceptance) as a foundation due to substantial evidence of the benefits of mindfulness in university students. However, subgroups within the university student population may respond differently to standard mindfulness instruction.

Indeed, emerging evidence suggests that mindfulness instruction may be experienced in unique ways by certain vulnerable populations, such as those with a history of non-suicidal self-injury (NSSI; self-injury without lethal intent) or attention-deficit/hyperactivity disorder (ADHD; neurodevelopmental disorder characterized by developmentally atypical levels of inattention and/or hyperactivity-impulsivity). Students with a history of engaging in NSSI comprise 10-39% of university students, while students with ADHD comprise 2-8% of university students. These subgroups of students tend to exhibit a vulnerability to university stressors and stand to incur important benefits from resilience-building strategies that are tailored to their needs.

However, students with history of NSSI or ADHD are predisposed to find standard mindfulness instruction challenging and/or inaccessible. Standard mindfulness instruction generally consists of a combination of formal and informal practice. Formal practices can be conceptualized as structured, sustained attentional guided activities in which mindfulness is practiced within an allotted period of time (e.g., sitting meditation, body scan), whereas informal practices are brief and unstructured, and focus on the experience of one's senses during routine activities (e.g., becoming aware of the feeling of water on one's hands while washing them). Formal practice often requires sustained attention on one's inner experience (i.e., thoughts and emotions) and bodily sensations. Existing difficulties with emotion regulation, self-criticism, and a potentially complex relationship with their body may render this common component of formal mindfulness practice challenging for students with a history of NSSI. For students with ADHD, the elevated level of attentional demand required for formal mindfulness practice may be particularly challenging (e.g., ADHD). Indeed, individuals with ADHD tend to report elevated attrition rates from mindfulness-based programs. If standard mindfulness programming is not properly adapted to individual differences, this may limit its accessibility to university students with a history of NSSI or ADHD.

Promising emerging evidence from our team finds that adolescents, who have difficulties with sustained attention, prefer informal mindfulness practice over formal practice. Specifically, students found the informal practices more accessible (more likely to use in future) than formal practices. This study is an important precursor to the proposed study, given that it provides reason to believe that students with ADHD, who also experience attention difficulties, might similarly find informal mindfulness more accessible. Similarly, a recent study by our team found that university students with a history of NSSI found informal mindfulness practice to be more acceptable than formal practice. Consistent with these exciting early results from our team, in a recent systematic review examining the unique benefits of informal mindfulness, it was concluded that informal practices may be more accessible and acceptable among those already experiencing difficulties with attention or emotion regulation. The need for additional studies exploring the potentially differential effectiveness of formal and informal mindfulness instruction among groups with unique intrapersonal needs was highlighted.

To investigate whether the response to and associated benefit of formal or informal mindfulness instruction differs between students with a history of NSSI or ADHD, the proposed study will use a randomized controlled design to investigate group differences in both the immediate response to, and long-term benefits of, formal versus informal mindfulness instruction. Specifically, the study will assess (1) satisfaction with each mindfulness instruction type quantitatively (through surveys) and qualitatively (through semi-structured interviews), (2) changes in mental health/well-being and educational outcomes over time, across groups (i.e., NSSI, ADHD, comparison) and conditions (i.e., formal, informal), and (3) whether the impact of the instruction (i.e., formal, informal, control) on these outcomes occurs as a function of changes in specific facets of mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Current student at McGill University or Concordia University
* 18-29 years old
* Either self-reported stress or self-reported ADHD or a self-reported history of engaging in NSSI on at least 5 separate days in the last year

Exclusion Criteria:

* Having a history of NSSI that does not fulfill the recency/frequency requirement

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Dispositional mindfulness | Weeks 1, 6, 10, and 18
  The 39-item Five Facets of Mindfulness Questionnaire (FFMQ) will be used to assess dispositional mindfulness. The FFMQ consists of five subscales, each reflecting one facet of mindfulness (acting with awareness, nonjudgmental acceptance, nonreactivity, observing, and describing). Items are rated on a 5-point Likert scale ranging from Never or very rarely true (1) to Very often or always true (5). Global or subscale sum scores may be calculated, whereby higher sum scores reflect greater levels of dispositional mindfulness (either globally or on that specific subscale). Dispositional mindfulness will be assessed across groups and conditions, as well as over time.

SECONDARY OUTCOMES:
Emotion regulation style | Weeks 1, 6, 10, and 18
  The 18-item Emotion Regulation Inventory (ERI) will be used to assess emotion regulation styles. The ERI consists of three subscales, each pertaining to one of three emotion regulation styles: integrative emotion regulation, suppressive emotion regulation, and dysregulated emotion regulation. All items are rated on a 5-point Likert scale ranging from Completely disagree (1) to Completely agree (5). Higher sum scores on the ERI subscales indicate greater levels of that specific ER style. Emotion regulation styles will be assessed across groups and conditions, as well as over time.
Psychological need satisfaction and frustration | Weeks 1, 6, 10, and 18
  The 24-item Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) will be used to assess satisfaction and frustration of the psychological needs for autonomy, relatedness, and competence. The BPNFS includes six, four-item subscales (autonomy satisfaction, autonomy frustration, relatedness satisfaction, relatedness frustration, competence satisfaction, and competence frustration), although its subscales may also be combined to create global measures of need satisfaction and need frustration. Items are rated on a 5-point Likert scale ranging from Completely disagree (1) to Completely agree (5). Higher sum scores indicate greater levels of need satisfaction/frustration globally or in that specific domain (i.e., autonomy, relatedness, competence). Psychological need satisfaction and frustration will be assessed across groups and conditions, as well as over time.
Stress | Weeks 1, 6, 10, and 18
  The 10-item Perceived Stress Scale will be used to assess perceived stress (PSS-10). Items are rated on a 5-point Likert scale ranging from Never (1) to Very often (5). A higher sum score indicates higher perceived stress. Stress will be assessed across groups and conditions, as well as over time.
Well-being | Weeks 1, 6, 10, and 18
  The 14-item Warwick-Edinburgh Mental Well-Being Scale will be used to assess well-being (WEMWBS). The WEMWBS is a unidimensional self-report questionnaire, with items related to various aspects of well-being including positive affect, satisfying interpersonal relationships, and positive functioning. Items are rated on a 5-point Likert scale ranging from None of the time (1) to All of the time (5) based on the extent to which each statement describes the respondent's experience over the last two weeks. A higher sum score indicates higher well-being. Well-being will be assessed across groups and conditions, as well as over time.
Academic engagement | Weeks 1, 6, 10, and 18
  The 9-item Utrecht Work Engagement Scale for Students will be used to assess academic engagement (UWES-S). The UWES-S is the student version of the most widely used measure to assess work engagement, the Utrecht Work Engagement Scale. The UWES-S assesses three aspects of academic engagement: vigor, dedication, and absorption. Items are rated on a 7-point Likert scale ranging from Never (1) to Always/every day (7). A higher mean score indicates higher academic engagement. Academic engagement will be assessed across groups and conditions, as well as over time.
Acceptability (as measured by the TFA questionnaire) | Weeks 6, 10, and 18
  The Theoretical Framework of Acceptability (TFA) Questionnaire will be used to assess participants' satisfaction with, and the acceptability of, their assigned intervention. This measure assesses the seven components of the TFA (affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy) which can help to identify characteristics of interventions that may be improved. The TFA Acceptability Questionnaire is adaptable and can be used to evaluate a variety of healthcare interventions (including mental healthcare). It consists of seven items, each pertaining to one of the components listed above, as well as an eighth item that assesses general acceptability. All items are rated on 5-point Likert scales. A higher mean score indicates higher acceptability. Acceptability will be assessed across groups and conditions, as well as over time.
Acceptability (as measured by the IMI) | Weeks 6, 10, and 18
  Subscales of the Intrinsic Motivation Inventory (IMI) will also be used to assess acceptability from a Self-Determination Theory perspective, as the IMI is intended to assess participants' subjective experience of a target activity in experimental research. For the purposes of this study, four subscales of this measure will be included: interest/enjoyment (5 items), perceived competence (5 items), perceived autonomy (6 items), and value/usefulness (7 items). All items are rated on a 7-point Likert scale ranging from Not at all true (1) to Very true (7). A higher mean score indicates higher acceptability. Acceptability will be assessed across groups and conditions, as well as over time.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Heath, Ph.D., Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Concordia University, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of findings, de-identified data will be uploaded to a public online repository (e.g., the McGill University Dataverse, the Open Science Framework [OSF]).